CLINICAL TRIAL: NCT00102154
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study of MK0928 in Healthy Adult Volunteers Participating in a 4-Hour Phase Advance Model of Transient Insomnia
Brief Title: An Investigational Drug Study in Healthy Adult Volunteers in a Model of Insomnia (0928-007)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-007; 2004_093
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0928, gaboxadol / Duration of Treatment: 10 months

SUMMARY:
A study to evaluate the safety and effectiveness of an investigational drug for insomnia (a sleep disorder).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are between the ages of 18 and 64

Exclusion Criteria:

* Adults who are diagnosed with insomnia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01

PRIMARY OUTCOMES:
4-hour advanced polysomnographic (PSG) recording session measuring wake time after sleep onset (WASO) and latency to persistent sleep (LPS); Safety and tolerability

SECONDARY OUTCOMES:
Daily sleep diary for visual analogue sleep quality and number of night awakenings (sNAW)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC